CLINICAL TRIAL: NCT05109741
Title: Internet-based Psychodynamic Therapy Compared to Behavioral Activation - a Randomized Controlled Trial
Acronym: ELSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Stockholm University (Other)
Responsible Party: Principal Investigator, Robert Johansson, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KIELSA1
Record Dates: First submitted 2021-10-27; First posted 2021-11-05 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Depression
Keywords: Psychotherapy; Psychodynamic therapy; Behavioral activation; Internet
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Internet-based Psychodynamic Therapy (Experimental): This is a 10-week treatment based on the psychodynamic SUBGAP model ("Seeing, Understanding, Breaking, and Guarding Against Patterns") by Farrell Silverberg (2005). The treatment has been evaluated in two previous randomized controlled trials.
  Silverberg, F. (2005). Make the leap: A practical guide to breaking the patterns that hold you back. Da Capo Press.
  Andersson, G., Paxling, B., Roch-Norlund, P., Östman, G., Norgren, A., Almlöv, J., ... & Silverberg, F. (2012). Internet-based psychodynamic versus cognitive behavioral guided self-help for generalized anxiety disorder: a randomized controlled trial. Psychotherapy and psychosomatics, 81(6), 344-355.
  Johansson, R., Ekbladh, S., Hebert, A., Lindström, M., Möller, S., Petitt, E., ... & Andersson, G. (2012). Psychodynamic guided self-help for adult depression through the internet: a randomised controlled trial. PloS one, 7(5), e38021.
  Interventions: Behavioral: Internet-based Psychodynamic Therapy
- Internet-based Behavioral Activation (Active Comparator): This 10-week treatment is based on the BATD-R ("Behavioral Activation Treatment for Depression - Revised") treatment by Lejuez and others (2011).
  Lejuez, C. W., Hopko, D. R., Acierno, R., Daughters, S. B., & Pagoto, S. L. (2011). Ten year revision of the brief behavioral activation treatment for depression: revised treatment manual. Behavior modification, 35(2), 111-161.
  Interventions: Behavioral: Internet-based Behavioral Activation
- Waiting-list (No Intervention): Participants will be in a 10-week waiting period.

INTERVENTIONS:
Behavioral: Internet-based Psychodynamic Therapy — Internet-based Psychodynamic Therapy based on the SUBGAP model developed by Farrell Silverberg
  Arms: Internet-based Psychodynamic Therapy
Behavioral: Internet-based Behavioral Activation — Internet-based Behavioral Activation based on the BATD-R model developed by Carl Lejuez and others.
  Arms: Internet-based Behavioral Activation

SUMMARY:
There are several treatment options for depression, including Internet-delivered psychotherapy. While a majority of this research is based on cognitive behavior therapy (ICBT), there are also several recent studies investigating Internet-delivered psychodynamic therapy (IPDT). Importantly though, these treatments have never been directly compared in a randomized controlled trial.

In this project, we aim to include 350 patients with depression randomized to ten weeks of IPDT (N=150), ICBT in the form of behavioral activation (N=150) or waiting list (N=50). After the end of the treatment period, patients on the waiting list will also be offered treatment. A secure web platform (KI eHealth Core Facility) will be used to provide treatment via the Internet.

Symptoms of depression will be measured weekly and the effect will be evaluated by comparing the change in the treatment groups with each other and with the change in the waiting list group. Treatment effects and predictors of treatment response will be examined.

In summary, this project is an important step in the continued evaluation of internet-based psychological treatments for depression.

DETAILED DESCRIPTION:
Depression is a widespread problem in Sweden and the world. The condition causes great suffering for the affected individual and his or her family, and involves major costs for society. There is promising support for psychological treatment of depression in the form of cognitive behavioural therapy and psychodynamic therapy, among others, also as self-help treatment in an internet-based format.

Internet psychodynamic therapy (IPDT) has shown significant effects in the treatment of both depression and anxiety disorders, but also in the treatment of somatic problems. The effects also appear to have improved from end of treatment to follow-up in most studies, with subjects largely completing the full treatment programme. In conclusion, the results for this form of treatment are very promising.

However, internet-based psychodynamic therapy for depression has never been compared with Internet-based CBT (ICBT) in a randomised controlled trial. This is not only an important issue from the perspective of comparing efficacy. Such a comparative study could also provide a basis for gathering information on predictors of treatment response. Based on the psychotherapy literature, there is reason to believe that different patients respond to different treatments. Thus, a comparative study between ICBT and IPDT may also provide a basis for answering the question "Which works for whom?".

In this project, we aim to include 350 patients with depression randomized to ten weeks of IPDT (N=150), ICBT in the form of behavioral activation (N=150) or waiting list (N=50). After the end of the treatment period, patients on the waiting list will also be offered treatment. A secure web platform (KI eHealth Core Facility) will be used to provide treatment via the Internet.

Symptoms of depression will be measured weekly and the effect will be evaluated by comparing the change in the treatment groups with each other and with the change in the waiting list group. Treatment effects and predictors of treatment response will be examined.

In summary, this project is an important step in the continued evaluation of internet-based psychological treatments for depression.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* A total score ≥10 on the PHQ-9

Exclusion Criteria:

* A score of >1 on the PHQ-9 item 9
* A total score >20 on the PHQ-9
* A psychological condition that might require other treatment (e.g., psychosis, suicidality, etc)
* Alcohol or substance addiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Baseline
  Self-report measure of symptoms of depression
Patient Health Questionnaire-9 (PHQ-9) | Post-treatment (10 weeks)
  Self-report measure of symptoms of depression
Patient Health Questionnaire-9 (PHQ-9) | 6-month follow-up
  Self-report measure of symptoms of depression
Patient Health Questionnaire-9 (PHQ-9) | 12-month follow-up
  Self-report measure of symptoms of depression

SECONDARY OUTCOMES:
General Anxiety Questionnaire-7 (GAD-7) | Baseline
  Self-report measure of symptoms of anxiety
General Anxiety Questionnaire-7 (GAD-7) | Post-treatment (10 weeks)
  Self-report measure of symptoms of anxiety
General Anxiety Questionnaire-7 (GAD-7) | 6-month follow-up
  Self-report measure of symptoms of anxiety
General Anxiety Questionnaire-7 (GAD-7) | 12-month follow-up
  Self-report measure of symptoms of anxiety
Brunnsviken Brief Quality of life scale (BBQ) | Baseline
  Self-report measure of quality of life
Brunnsviken Brief Quality of life scale (BBQ) | Post-treatment (10 weeks)
  Self-report measure of quality of life
Brunnsviken Brief Quality of life scale (BBQ) | 6-month follow-up
  Self-report measure of quality of life
Brunnsviken Brief Quality of life scale (BBQ) | 12-month follow-up
  Self-report measure of quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Robert Johansson, PhD, Principal Investigator — Stockholm University and Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No